CLINICAL TRIAL: NCT02257437
Title: Acceptability of a Locally-Produced Multiple Micronutrient-Fortified Lipid-Based Nutrient Supplement (LNS) for Children Under Two Years in Cambodia
Brief Title: Acceptability of a Multiple Micronutrient-Fortified Lipid-Based Nutrient Supplement for Children Under Two in Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement, Cambodia (Other Government)
Collaborators: UNICEF (Other); Department of Fisheries Post-harvest Technologies and Quality Control (Other)
Responsible Party: Principal Investigator, Bindi Borg, PhD Candidate, University of Sydney
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LNS-CAMB-INFANTS
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Child Malnutrition
Keywords: Ready-to-use supplementary food (RUSF); Lipid-based nutrient supplement (LNS); Multiple micronutrients (MMN); Complementary feeding; Home fortification; Acceptability; Infant and young child feeding (IYCF); Cambodia; Cross-over studies
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Hypoxanthine Phosphoribosyltransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LNS + borbor (Experimental): Lipid-based nutrient supplement (LNS) added to borbor
  Interventions: Dietary Supplement: LNS snack; Dietary Supplement: Corn-soy blend ++ (CSB++); Dietary Supplement: Sprinkles; Dietary Supplement: LNS + borbor
- Corn-soy blend ++ (CSB++) (Active Comparator): CSB++ porridge
  Interventions: Dietary Supplement: LNS snack; Dietary Supplement: Corn-soy blend ++ (CSB++); Dietary Supplement: Sprinkles; Dietary Supplement: LNS + borbor
- Sprinkles (Active Comparator): Sprinkles added to borbor
  Interventions: Dietary Supplement: LNS snack; Dietary Supplement: Corn-soy blend ++ (CSB++); Dietary Supplement: Sprinkles; Dietary Supplement: LNS + borbor
- LNS snack (Active Comparator): LNS eaten as snack
  Interventions: Dietary Supplement: LNS snack; Dietary Supplement: Corn-soy blend ++ (CSB++); Dietary Supplement: Sprinkles; Dietary Supplement: LNS + borbor

INTERVENTIONS:
Dietary Supplement: LNS snack — Compact, paste-filled wafer snack containing fish, rice, soy, mungbeans, oil, sugar and multiple micronutrients.
Dietary Supplement: Corn-soy blend ++ (CSB++) — Blended flour containing soy, corn, milk powder, oil, sugar and multiple micronutrients.
  Other Names: Supercereal Plus
Dietary Supplement: Sprinkles — Multiple micronutrient powder packaged in sachet added to borbor (traditional white rice porridge).
Dietary Supplement: LNS + borbor — Compact, paste-filled wafer snack containing fish, rice, soy, mungbeans, oil, sugar and multiple micronutrients added to borbor (traditional white rice porridge).

SUMMARY:
The purpose of this trial is to evaluate the acceptability of the LNS to women and their children aged 12-17 months in comparison to Corn Soy Blend++, and Sprinkles added to borbor (white rice porridge, which is the traditional weaning food in Cambodia). Acceptability will be assessed through a sensory test for caregivers, and by measuring children's consumption.

DETAILED DESCRIPTION:
BACKGROUND:

In Cambodia, progress in combatting malnutrition has stalled. In 2010, 40% of all children under five (and 49% of 4-5 year-olds) were stunted, 11% were wasted, and 28% were underweight, indicating, respectively, chronic and acute malnutrition, and a combination of the two. Stunting is partially attributed to poor complementary feeding, which remains inadequate for achieving growth outcomes and micronutrient status.

Malnutrition can be prevented and treated with supplementary foods. These foods usually contain a source of protein and lipids such as powered milk, soy or peanuts, and multiple micronutrients. They can be prepared as a fortified blended product, such as Corn-Soy Blend++ (CSB++), that is mixed with water to make a porridge, or ready-to-use supplementary foods (RUSFs). The latter are usually lipid-based nutrient supplements (LNSs) which are often pastes such as the peanut-based Plumpy'Nut™. These energy-dense supplementary foods contain both macro and micronutrients and are used to prevent and treat malnutrition by promoting improved linear growth, weight gain and micronutrient status among children. Until recently, prevention of malnutrition has relied on fortified blended products. The new RUSFs are also proving effective, as they are higher energy and have a longer shelf life, and since they require no preparation, are convenient. Another common nutrition intervention is multiple micronutrient supplements such as Sprinkles. These are individually-packed powders that can be added to food. However, micronutrients are more likely to achieve growth outcomes when they are combined with energy, for example, in lipid-based nutrient supplements and there is no evidence that micronutrient powders alone contribute to growth.

Until June 2014, the United Nations World Food Program (WFP) used CSB++ (now called Supercereal Plus) to prevent malnutrition in Cambodia. Sprinkles are also being distributed, though not widely, to prevent micronutrient deficiencies. These products that have been recently or are currently used are relatively expensive to procure and ship to Cambodia and in the case of Sprinkles, are not as effective as foods that contain macronutrients. Moreover, CSB++ was not very well accepted in practice, and WFP has phased it out. Therefore, UNICEF and the Cambodian Ministry of Health are looking for a locally-produced product containing macro and micronutrients to prevent malnutrition in Cambodia. Locally-produced products are more likely to be acceptable and cheaper than imported products.

Regardless of how effective a product may be, it is vital to determine its acceptability in a given setting, in other words, will a child eat the product and will a caregiver feed it to them. Acceptability to children can be measured by how much they eat and how readily, while acceptability to caregivers is measured in terms of their sensory perception of the food, that is, of the smell, colour, and taste.

TRIAL DESIGN AND METHODOLOGY:

Therefore, this trial will evaluate the acceptability of the LNS to women and their children aged 9-23 months in comparison to CSB++, Sprinkles added to borbor.

The trial is a cluster randomised, incomplete block, 4 x 4 crossover design that aims to establish the superiority (i.e. the greater acceptability) of the novel LNS (as a snack or mixed with borbor), in comparison to CSB++, and Sprinkles added to borbor. The allocation ratio is 1:1. The study will take place in two parts over two weeks:

1. Substudy 1: Acceptability by children, three days x four foods for a total of 12 days
2. Substudy 2: Acceptability by mothers, 13th day

The study will be conducted in peri-urban Phnom Penh. The study will be conducted in four test-feeding sites such as pagodas or health centres. Participants will be recruited for convenience from villages close to the four sites. The four test-feeding sites will be randomly allocated to begin on one of the foods. All children in a given site will be eating the same food at the same time for three consecutive days.

Upon consent and enrolment, baseline data will be collected from the participants. This will include demographics, morbidity, anthropometry (weight, height, mid-upper arm circumference), and dietary data (breastfeeding, food frequency and dietary diversity).

Mothers will be asked to bring their child to their designated test-feeding site for the following 12 days. They will be asked not to feed their child for the preceding hour, if possible. The same food will be given three days in a row, to allow averaging of results and reduce the effect of chance findings.

Children will receive the four foods, namely, the LNS added to borbor, CSB++ porridge, Sprinkles added to borbor, and the LNS snack, for three days each over twelve days. Children in each group will taste each food in a different sequence (to balance for carry-over effects). The mothers will be asked to feed their child for 15 minutes or until the child refuses to eat any more. The amount of food consumed will be measured each time the child eats. Each mother will be asked to assess how she thinks her child liked the food, taking into account the amount eaten and the child's reactions and emotional state during feeding.

On the 13th day, mothers will be asked to come to the test-feeding site, alone if possible, to rank the foods. For the sensory test, the foods will be presented one at a time. No weighing is necessary and mothers will not be expected to eat a whole cup. Between foods, the mother will be asked to rinse her mouth out with water. Mothers will rate each food with respect to colour, smell, taste, preparation process, and their overall opinion. The foods will then be presented at the same time and mothers will then be asked to rank them. Finally, on the 14th day, a smaller number of mothers (8-12) from each site will be asked to stay for a focus group discussion related to infant feeding practices and reasons for preference ranking.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9-23 months and their caregivers
* Have been eating solids for at least three months
* Singletons
* Normally nourished or only moderately malnourished (MUAC >115mm, WHZ score >-3)
* Healthy (no ill-health in past three days)
* No known food intolerances
* Have not been using Sprinkles, CSB++ or similar supplementary foods or supplements
* Informed signed consent of mother
* Mothers are healthy

Exclusion Criteria:

* Children <9 months or >23mths
* Not yet eating solid food for at least three months
* Twins/multiples
* Severely malnourished (MUAC< 115mm, WHZ score<3, bipedal pitting oedema).
* Oedema and/or any medical complications at recruitment or illness requiring referral, or any ill health in past three days.
* Known intolerances
* Children enrolled in Sprinkles, CSB++ or similar program
* No informed signed consent of caregiver
* Medical complications or illness requiring referral at time of recruitment or previous two weeks

Ages: 9 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Child's consumption | Within 15 minutes
  How much of a given food the children consume

SECONDARY OUTCOMES:
Child's preference | 3 days
  Mothers' assessment of their child's ranked preference for the food
Mother's ranking | 1 session
  Mother's ranked preference for the food

CONTACTS AND LOCATIONS:
Overall Officials: Frank T Wieringa, MD, PhD, Study Director — IRD; Bindi Borg, PhD student, Principal Investigator — University of Sydney
Locations (1):
- IRD Cambodia, Phnom Penh, Cambodia

REFERENCES:
- [Derived] Borg B, Mihrshahi S, Griffin M, Chamnan C, Laillou A, Wieringa FT. Crossover trial to test the acceptability of a locally produced lipid-based nutrient supplement (LNS) for children under 2 years in Cambodia: a study protocol. BMJ Open. 2017 Sep 6;7(9):e015958. doi: 10.1136/bmjopen-2017-015958. PMID 28882910